CLINICAL TRIAL: NCT02532413
Title: Comparison of Antiviral Efficacy of Entecavir Monotherapy and Combination Treatment With Poly IC for Chronic Hepatitis B
Brief Title: Antiviral Efficacy of the Combination Treatment With Poly IC and Entecavir for Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xin Zheng, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81461130019C5
Record Dates: First submitted 2015-07-24; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Poly I-C; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HBeAg(+):Poly IC+Entecavir (Experimental): 45 subjects(HBeAg-positive chronic hepatitis B). Combination therapy will last 24 weeks from 0 week.
  Drug: Entecavir 0.5mg, P.O.,qd, duration:48 weeks. Drug: PolyIC 2mg,im,qod,duration:from 0 week to 24th week
  Interventions: Drug: Poly IC; Drug: Entecavir
- HBeAg(+):Entecavir (Active Comparator): 45 subjects(HBeAg-positive chronic hepatitis B). Drug: Entecavir 0.5mg, P.O.,qd, duration:48 weeks.
  Interventions: Drug: Entecavir
- HBeAg(-):Poly IC+Entecavir (Experimental): 45 subjects(HBeAg-negative chronic hepatitis B). Combination treatment will last 24 weeks from 0 week.
  Drug: Enticavir 0.5mg, P.O.,qd, duration:48 weeks. Drug: PolyIC 2mg,im,qod,duration:from 0 week to 24th week
  Interventions: Drug: Poly IC; Drug: Entecavir
- HBeAg(-):Entecavir (Active Comparator): 45 subjects(HBeAg-negative chronic hepatitis B). Drug: Entecavir 0.5mg, P.O.,qd, duration:48 weeks.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Poly IC — Poly IC can induce innate immune responses.It may enhance the antiviral efficacy of Entecavir.
  Other Names: Polyinosinic-polycytidylic acid injection
  Arms: HBeAg(+):Poly IC+Entecavir; HBeAg(-):Poly IC+Entecavir
Drug: Entecavir — Entecavir can inhibit the replication of HBV.
  Other Names: Leiyide

SUMMARY:
The purpose of this study is to investigate antiviral efficacy of the combination treatment with Poly IC and Entecavir and compare with the efficacy of Entecavir mono-therapy for chronic hepatitis B.

DETAILED DESCRIPTION:
In this study, the patients with chronic HBV infection will be divided into two groups: HBeAg (+) and HBeAg (-) group. Each group will be divided into two subgroups, which are treated with combination treatment of Entecavir and Poly IC and Entecavir monotherapy respectively. All the patients will be followed up for one year. From this study, the investigators want to study if Poly IC can enhance antiviral efficacy of Entecavir for chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months.
* Having been treated wit Entecavir and the level of HBV DNA is under 1000 copies/ml.
* ALT ≤10×ULN， TB <2ULN .

Exclusion Criteria:

* Previous antiviral treatment for HBV.
* Co infection of HIV, HCV, HEV, HAV, or HAV.
* Evidence of hepatic carcinoma.
* Evidence of autoimmune disease.
* Evidence of thyroid disease.
* History of mental sickness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with HBsAg serological response | at week 48 of treatment
  The proportion of patients who achieve HBsAg serological response as assessed by the rate of HBsAg seroconversion.

SECONDARY OUTCOMES:
Changes in serum HBV DNA levels | at week 4，12，24，36，48，72，96 of treatment
  Changes in serum HBV DNA levels during 48 weeks of treatment
Biochemical Response （the serum levels of ALT and AST） Biochemical Response | at week 1，2，4，8，12，16，20，24，36，48，72，96 of treatment
  Biochemical response as assessed by the serum levels of ALT, AST, TB, etc.
Proportion of patients with HBeAg serological response | at week 48 of treatment
  The proportion of patients who achieve HBeAg serological response as assessed by the rate of HBeAg loss or HBeAg seroconversion.

CONTACTS AND LOCATIONS:
Overall Officials: Liang D Yang, M.D., Study Chair — Huanzhong University of Science and Technology
Locations (1):
- Department of Infectious Disease of Wu Han Union Hospital, Wuhan, Hubei, China